CLINICAL TRIAL: NCT02104726
Title: Prospective Randomized-Controlled Two-Arm Study of "Blind" vs. Fluoroscopy-Guided Steroid Injections for Knee Osteoarthritis
Brief Title: "Blind" vs. Fluoroscopy-Guided Steroid Injections for Knee Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00026934
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (2):
- Blind Steroid Injection (Active Comparator): Blind Steroid Injection for patients with OA deemed qualified for it clinically
  Interventions: Other: Blind Steroid Injection
- Fluoroscopy guided steroid injection (Active Comparator): Fluoroscopy guided Steroid Injection for patients with OA deemed qualified for it clinically. We want to see which one is better.
  Interventions: Other: Fluoroscopy guided steroid injection

INTERVENTIONS:
Other: Fluoroscopy guided steroid injection — We want to compare if there is a difference between the two arms, with the assumption that with fluoroscopy will deliver the steroid more accurately and see better outcomes.
  Arms: Fluoroscopy guided steroid injection
Other: Blind Steroid Injection — Want to compare it to fluoroscopy guided, with assumption that it will be less effective in reducing pain
  Arms: Blind Steroid Injection

SUMMARY:
To compare relative efficacy of intraarticular steroid injection using anatomic landmarks vs. fluoroscopy guided technique in decreasing knee osteoarthritis pain 1 month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

- Adults with knee OA clinically deemed to qualify for steroid injection

Exclusion Criteria:

- Children Non-English Speakers Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (pain) | 1 month
  Decrease in pain from baseline at one month